CLINICAL TRIAL: NCT01655459
Title: Evaluation of the LMA Position Using Ultrasound in Pediatric Patients
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2011-0800
Record Dates: First submitted 2012-07-24; First posted 2012-08-01 (Estimated); Last update posted 2012-08-01 (Estimated); Status verified 2012-07

CONDITIONS: Infraumbilical Surgeries
Keywords: ultrasound, LMA, fiberoptic bronchoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Ultrasound exam of upper airway: Following Internal Review Board approval(4-2011-0800) and written informed consent, total 100 patients(ASA I and II children aged 1 month to 6years) undergoing infra-umblicular urologic surgeries were included in the study. Children with upper respiratory tract infection, restricted mouth opening, congenital heart disease and those at risk for aspiration were excluded.
  Interventions: Procedure: Ultrasound exam of upper airway

INTERVENTIONS:
Procedure: Ultrasound exam of upper airway — LMA-position was evaluated with fiberoptic laryngoscopy. The ultrasound findings of pre- and post-LMA were compared.

SUMMARY:
Introduction: Although the LMA insertion is not difficult and majority of the cases with LMA fare well in ventilation, the FOB assessment demonstrates a high incidence of LMA malpositioning. The LMA must be seated at the laryngeal inlet with the occlusion of esophageal inlet by the inflated tip. When we meet the signs of LMA malposition, we then reinsert the LMA. The laryngoscopic grading of Rowbottom et al. is commonly used for LMA position, but the rotated degree of LMA was not considered in that grading. We hypothesized that the LMA can affect the position of the arytenoids/thyroid cartilages and it may be detected on ultrasound. This study was designed to assess the predictability of the rotated LMA according to the position change of arytenoids/thyroid cartilages using ultrasound.

Methods: Children, aged 1 ms - 6 years, undergoing infraumbilical surgery were enrolled to this study. Ultrasound was performed on supraglottic and vocal cords area before and after LMA insertion. Transverse images were obtained on end-expiratory phase. LMA-position was evaluated with Bonfils fiberscopy. Position grading was made as usual. If grade >3 was showed, LMA was repositioned while fiberscopic watching. If the face of LMA was rotated to one-side, the LMA was rotated to the opposite side a little. The ultrasound findings of pre- and post-LMA were compared. On fiberscopic images, conventional LMA grade and the degree of rotation were measured.

ELIGIBILITY:
Inclusion Criteria:

* Aged 1 ms - 6 years,
* undergoing infraumbilical surgery

Exclusion Criteria:

* coagulopathy
* pathologic lesions on neck or upper airway
* mallampati class III or IV
* difficult airway past history
* high risk group of aspiration pneumonitis

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Following Internal Review Board approval(4-2011-0800) and written informed consent, total 100 patients(ASA I and II children aged 1 month to 6years) undergoing infra-umblicular urologic surgeries were included in the study. Children with upper respiratory tract infection, restricted mouth opening, congenital heart disease and those at risk for aspiration were excluded.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2012-01; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
changes of Ultrasound image of upper airway after Fiberoptic bronchoscopic grade of LMA insertion. | After the induction of general anesthesia, ultasound image was gained before and after the LMA insertion. Fiberoptic bronchoscpy was done after the LMA insertion.